CLINICAL TRIAL: NCT07190417
Title: Evaluation of Physiological Effects Induced by Low Level Light Irradiation on the Acupoints of the Hand
Acronym: Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YM109166F
Record Dates: First submitted 2025-03-04; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2024-05

CONDITIONS: Insomnia; Anxiety; Acupuncture; Low-level Laser Therapy
Keywords: Insomnia; Anxiety; Acupuncture; Acupoint Stimulation; Low-Level Laser Therapy (LLLT); Heart Rate Variability (HRV); Meridian Energy; Traditional Chinese Medicine (TCM)
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders | interventions — Lasers; Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Preliminary experiment on low-energy laser acupuncture for insomnia (healthy subjects, single-blind) (Sham Comparator): Objective:
  To evaluate the effectiveness of low-energy LED therapy on acupoints in treating insomnia, considering Fitzpatrick skin type variations.
  Methods:
  90 participants (Fitzpatrick types I-VI) from National Yang-Ming Chiao Tung University will be recruited.
  Participants will receive either low-energy LED or sham therapy for 25 minutes, twice, in a controlled environment.
  Heart rate variability, meridian energy, and light penetration will be measured before, during, and after the intervention.
  Note: This version removes unnecessary details about the time of day, temperature, and eye safety. It focuses on the core elements of the study: the intervention, the participants, the measurements, and the overall objective.
  Interventions: Other: LEDs and laser light
- Preliminary experiment on the use of low-energy LED for acupuncture for insomnia (Double-blind) (Sham Comparator): This experiment is similar to Experiment A, but the sham light intervention will use a sham device. The design will be double-blind.
  Experiment personnel (B) will randomly assign participants to wear either the low-energy LED device or the sham device. Experiment personnel (A) will assist participants in wearing the devices and measuring signals. Prior to the completion of the experiment, personnel (A) will not be aware of which device (LED or sham) is actually emitting light (the near-infrared light from the LED is difficult to see even with the naked eye after scattering). The low-energy LED device and the sham device will have identical indicator lights, operating cycles, and sound indicators.
  Interventions: Other: LEDs and laser light
- To investigate how light from LEDs and lasers penetrates different skin types. (Experimental): This study will investigate how light from LEDs and lasers penetrates different skin types.
  Participants:
  90 participants (Fitzpatrick Skin Types I-VI) will be recruited from National Yang-Ming Chiao Tung University.
  60 participants will be from previous experiments, and 30 from international students.
  Procedure:
  Categorize participants into six groups based on Fitzpatrick skin type. Measure initial light power of the LED and laser sources. Mark a target point on the participant's earlobe or ear cartilage. Measure the thickness of the earlobe/cartilage. Measure light power after penetrating through the earlobe/cartilage. Calculate light power reduction (attenuation) for LED and laser interventions. Analyze light transmission percentages across Fitzpatrick skin types to assess LED light penetration suitability.
  Goal: To determine if light penetration is affected by skin color.
  Interventions: Other: LEDs and laser light

INTERVENTIONS:
Other: LEDs and laser light — Experiment 1：Measure the heart rate parameters before, during, and after laser acupuncture or LED light therapy within a 25-minute experimental period, and observe the changes in the subjects' meridian energy before and after the treatment, followed by analysis. Acupoint selections mainly include Daling, Neiguan, and Shenmen.
  Experiment 2：randomly assigns subjects to wear either a low-energy LED device or a sham device. The indicators, duty cycles, and sounds of the low-energy LED device and the sham device are all the same.
  Experiment 3：Place light sources of different wavelengths on the earlobes or auricles of subjects with different skin tones. By observing the changes in light power before and after, the investigators can infer the effects of skin tone on light attenuation and transmission of light sources with different wavelengths.
  Other Names: LED; Laser therapy; laser acupuncture

SUMMARY:
The goal of this clinical trial is to determine if low-level laser therapy (LLLT) and LED-based low-level light therapy (LLLT) are effective in inducing relaxation and improving sleep quality and anxiety levels in individuals with insomnia. It aims to evaluate the potential of both light sources to elicit comparable physiological changes in relation to acupoint stimulation.

The main questions this trial aims to answer are:

Does exposure to low-level laser or LED light therapy on specific acupoints associated with insomnia result in similar changes in heart rate variability and meridian energy? How does skin pigmentation affect the penetration of different wavelength light sources used in LLLT? Primary hypothesis 1: Low-level LED light therapy is comparable to laser therapy in terms of effectiveness.

Primary hypothesis 2: With proper design, both treatments will elicit similar changes in meridian energy and heart rate variability.

Researchers will compare the effects of low-level laser and LED light therapy on 60 participants, divided into two groups: 30 healthy participants receiving either low-level laser/sham laser or low-level LED/sham LED light exposure and 30 participants with brown to black skin tones receiving different LED and laser specifications.

Participants will:

Undergo either low-level laser/sham laser or low-level LED/sham LED light exposure on specific acupoints.

Have their heart rate variability and meridian energy levels measured before and after the intervention.

Have their skin pigmentation measured to assess light penetration with various wavelengths.

This study seeks to establish a stronger link between acupoint stimulation, light therapy, and sleep neuroscience, potentially offering an alternative therapeutic approach for insomnia that complements existing pharmacological interventions.

DETAILED DESCRIPTION:
Research Background： In recent years, acupuncture has emerged as a promising therapeutic approach for improving sleep quality in menopausal women, particularly in addressing the challenging aspect of deepening sleep. This has led to an increased focus on acupunctural treatments, including acupoint stimulation, as a potential solution for insomnia. However, with increasingly stringent medical regulations, even non-invasive low-level laser therapy, despite its significantly safer profile compared to traditional acupuncture needles, faces substantial regulatory hurdles.

Meanwhile, novel LED technology presents a compelling alternative to lasers. Compared to lasers of equivalent power, LEDs boast lower costs, energy consumption, and operating temperatures without compromising therapeutic efficacy. This makes LED-based low-level light therapy (LLLT) a highly promising approach, especially for applications where diverse medical needs are present, such as in organizations like NASA.

This study is a preliminary investigation into the application of acupoint light therapy within the realm of Traditional Chinese Medicine (TCM) for managing insomnia and anxiety. The objective is to evaluate the potential of both low-level laser therapy and low-level LED light therapy, under similar power and wavelength conditions, to induce comparable physiological changes and consequently improve sleep quality and alleviate anxiety.

Specifically, this research will examine whether exposure to either light source results in similar relaxation effects by analyzing relevant physiological indicators like heart rate variability parameters and conductive meridian (Jingluo) parameters - a measure of electrical resistance along meridians. Furthermore, this study will address the understudied influence of skin pigmentation on LLLT by conducting optical experiments to determine the penetration depth of light sources with varying wavelengths through different skin types. This will contribute to a more comprehensive understanding of the application of LLLT in acupoint stimulation.

Research Objectives:

Investigate the effects of low-level laser and LED light therapy on acupoints associated with insomnia in the hands, using heart rate variability parameters and conductive meridian resistance (Jingluo) measurements as assessment tools.

Clarify the influence of skin pigmentation on the propagation of low-level laser and LED light by using a light power meter to quantify the difference in light transmission through darker and lighter skin types for various wavelengths.

Hypothesis:

Low-level LED light therapy is comparable to laser therapy in terms of its effectiveness. With proper design, both treatments will elicit similar changes in meridian energy and heart rate variability.

Data and Methods:

A total of 90 participants will be recruited for this study, divided into two groups:

Group 1: Consists of 30 healthy participants who will undergo either low-level laser/sham laser or low-level LED/sham LED light exposure. Changes in meridian energy and heart rate variability will be assessed after the intervention. Participants in this group will also be required to undergo pre- and post-light exposure measurements using different LED and laser specifications.

Group 2: Includes 30 participants with skin tones ranging from brown to black, categorized using the Fitzpatrick skin type scale. They will also undergo pre- and post-light exposure measurements using different LED and laser specifications.

Expected Results:

This study anticipates observing changes in meridian resistance and heart rate variability parameters following the application of low-level light stimulation to acupoints. By evaluating the penetration of light sources of various wavelengths through different human tissues, the study aims to establish a stronger link between LLLT and physiological indicators related to relaxation.

Significance:

This research aims to create a stronger connection between the practices of TCM acupoint stimulation, light therapy, and sleep neuroscience. The findings have the potential to provide an alternative therapeutic option for individuals suffering from insomnia, complementing existing pharmacologic interventions.

ELIGIBILITY:
Inclusion Criteria:

1. No use of sleeping pills within the past 3 months.
2. Pittsburgh Sleep Quality Index (PSQI) < 5 points.
3. Body Mass Index (BMI): 18.5 < BMI < 30.
4. Blood pressure: within normal range (<140 mmHg/90 mmHg).
5. Individuals with regular wake-sleep times: bedtime between 22:00 and 02:00.

Exclusion Criteria:

1. Individuals with insomnia and other sleep disorders.
2. Exclude those currently taking medications.
3. Individuals with cardiovascular diseases, cancer, psychiatric disorders, kidney diseases, diabetes, chronic illnesses, and physical discomfort.
4. Exclude individuals with addictions to smoking, alcohol, caffeine, and drugs.
5. Individuals with light sensitive skin.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Heart rate variability of Healthy Participant during Low-Energy LED Therapy | Measure three times: before, during, and after, each lasting 5 minutes
  Heart rate variability is measured by using Wegene Electrocardiogram Recorder (Medical Device License No. 004896 of the Ministry of Health): Developed by National Yang-Ming University and in cooperation with Wegene Technology, this handheld heart rate measurement system allows users to measure heart rate variability parameters in a relaxed manner and reflect the main parameters on the dashboard in real time. The primary unit of measure for heart rate variability (HRV). HRV reflects the variation in time between consecutive heartbeats(bpm), and this variation is typically very small, measured in milliseconds. HRV parameters includes Total Power, TP [ln(ms²)], Standard deviation of Normal to Normal R Wave, SDNN(ms²), High Frequency, HF [ln(ms²)], Low Frequency, LF [ln(ms²)], Very Low Frequency, VLF [ln(ms²)], percentage of HF(%), percentage of LF(%), LF/HF ratio.

SECONDARY OUTCOMES:
Meridian Energy Measurement of Healthy Participant during Low-Energy LED Therapy. | Measure two times: before and after, each lasting for 6 minutes
  A spring-loaded probe, is moistened with 5% saline and, after sterilization, applied sequentially to the 24 Yuan acupoints. After 2-3 seconds of 12 g/cm2 pressure for each point, the device is automatically interrupted, and the average value is recorded on a computerized system. In Meridian Energy Analysis (MEA), the primary unit of measure is electrical conductance, typically expressed in microamperes (μA). This measurement reflects the flow of electrical current through the meridian pathways, which can measure the vital energy (Qi) in traditional Chinese medicine. The MEA device used in the investigation is the Meridian Energy Analysis Device (MEAD). It uses a small electrical current (200 μA) to measure the Qi of the 24 pathways and their associated energy levels.

OTHER OUTCOMES:
To investigate how light from LEDs and lasers penetrates different skin types. | The experiment takes about 15 seconds for measuring and recording each light source, total time duration needed for each participants is 30 minutes.
  The difference in the transmission ratio of each wavelength among groups is measured by using Japan's SANWA LP10 optical power meter, unit used is 40mW (milliwatts). The rate from the power meter(40mW) is measure before and after the LED or lasers light are applied. The applicability of LED transmission are observed by calculating their attenuation ratio(%).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Brain Science, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No